CLINICAL TRIAL: NCT05551247
Title: A Prospective, Single-arm, Multicenter Clinical Trial of Envafolimab Combined With Recombinant Human Endostatin (Endostatin) in the Treatment of Recurrent or Metastatic MSS-type Colorectal Cancer
Brief Title: Envafolimab Combined With Endostatin in Recurrent or Metastatic MSS-type Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: No.XJTU1AF2022LSK-0076
Record Dates: First submitted 2022-05-31; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — envafolimab; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab plus recombinant human endostatin (endostatin) (Experimental): Envafolimab:300mg,sc,d3,Q3W; endostatin:210mg,civ,d1-3,Q3W.
  Interventions: Drug: Envafolimab; Drug: recombinant human endostatin (endostatin)

INTERVENTIONS:
Drug: Envafolimab — 300mg,sc,d3,Q3W;
Drug: recombinant human endostatin (endostatin) — 210mg,civ,d1-3,Q3W

SUMMARY:
The objective is to investigate the efficacy and safety of envafolimab combined with recombinant human endostatin (endostatin) in the treatment of MSS-type colorectal cancer patients with recurrence or metastasis after failure of second-line standard therapy.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, single-arm clinical study. That is, eligible colorectal cancer patients, after signing the informed consent form, are screened into the group, and will receive continuous intravenous infusion of envafolimab (envafolimab) combined with recombinant human endostatin (endostatin) until the disease. Progressive or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent form, and had good compliance;
* 18-75 years；
* ECOG 0-1；
* life expectancy of at least 3 months；
* Pathological specimens can be provided for biomarker detection
* Patients with recurrent or metastatic advanced MSS-type colorectal adenocarcinoma diagnosed by pathology and histology, and who are judged by the doctor to be suitable for receiving the nvolimab combined with recombinant human endostatin (endostatin) in this study.
* Previously received second-line standard systemic therapy (chemotherapy cycle at least ≥3 cycles), including fluorouracil or its derivatives, oxaliplatin, irinotecan and bevacizumab treatment, disease progression during or after treatment or Relapse, and have not received immune checkpoint inhibitor therapy before; Note: Patients who have received one regimen of adjuvant or neoadjuvant chemotherapy can be enrolled if they relapse > 6 months after the end of chemotherapy;
* Patients with MSS/pMMR type detected by PCR or IHC in the central laboratory;
* Patients with at least one measurable lesion according to RECIST 1.1, the efficacy evaluation standard for solid tumors, that is, in CT or MRI detection, the longest diameter of a single lesion is ≥10mm, or the lymph node is pathologically enlarged, and a single lymph node CT scan has a short diameter ≥15mm;
* Satisfactory main organ function，laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count（ANC） ≥1.5×109/L, platelet count（PLT） ≥80×109/L, Serum creatinine（CR）≤1.5 upper normal limitation (UNL)，total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; left ventricular ejection fraction (LVEF) ≥ 50%; thyroid stimulating hormone (TSH) within the normal range Within: if the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* Subjects of childbearing potential must use an appropriate method of contraception during the study period and within 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects

Exclusion Criteria:

* Suffered from other malignant tumors within 3 years before the start of treatment in this study;
* The pathological indication is mucinous adenocarcinoma and other special pathological types;
* Grade ≥1 unresolved toxicities (according to the most recent version of the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE]) due to any prior therapy, excluding alopecia and fatigue; neurotoxicity was Recovery to ≤ grade 1 or baseline before the group;
* Subjects with any severe and/or uncontrolled disease ；
* Poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L) ；
* Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment; or had a long-term unhealed wound or fracture；
* Serious arterial/venous thrombotic event within 6 months prior to initiation of study treatment ；
* Previously received drug therapy against PD-1, PD-L1 and other related immune checkpoints ；
* Participating in or participating in other clinical investigators within 4 weeks prior to the start of the study ；
* Allergic to the active ingredients or excipients of the study drug ；
* Unsuitable for the study or other chemotherapy determined by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2023-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
ORR | From Baseline to disease progress, up to 24 months
  Objective response rate

SECONDARY OUTCOMES:
PFS | From Baseline to primary completion date, about 2 years
  Progression Free Survival
OS | From Baseline to primary completion date, about 2 years
  Overall Survival
DCR | From Baseline to primary completion date, about 2 years
  Disease Control Rate
DOR | From Baseline to primary completion date, about 2 years
  Duration of Response
SAE | From Baseline to primary completion date, about 2 years
  severity Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Enxiao Li, Study Director — First Affiliated Hospital of Xian Jiaotong University

IPD SHARING:
Plan to Share IPD: No